CLINICAL TRIAL: NCT00260390
Title: The Efficacy of Testosterone Replacement in Treating Middle-Aged Hypogonadal Men With Dysthymia: Parallel Group, Double Blind Randomized Trial
Brief Title: Testosterone Replacement in Middle-Aged Hypogonadal Men With Dysthymia: Parallel Group, Double Blind Randomized Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-04-3222-GO-CTIL
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-10

CONDITIONS: Dysthymic Disorder
Keywords: Dysthymic Disorder; HPG hypofunctioning; Testosterone replacement
MeSH Terms: conditions — Dysthymic Disorder | interventions — Methyltestosterone

INTERVENTIONS:
Drug: Testoviron

SUMMARY:
Growing evidence supports the notion that Late-onset Dysthymic disorder in middle aged men may be associated with age-related HPG hypofunctioning. In this study we seek to examine the efficacy of Testosterone replacement for this condition.

Hypothesis:

Testosterone replacement will be more effective than placebo, in treating men with late onset Dysthymic Disorder and hypo-gonadism.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age 40-80 years.
2. Diagnosed with hypogonadism (total T level below 350 ng/dl), but not previously treated.
3. Diagnosis of Dysthymic disorder with onset after age 40.
4. PSA < 4.0.
5. Normal digital exam of the prostate in the preceding 1 year.
6. For subjects currently taking an antidepressant: Current antidepressant treatment last 6 weeks or longer, with decent dose and with no remission (or with partial remission only HAM-D > 12).
7. Able to give informed consent.

Exclusion Criteria:

1. Acute, severe, or unstable prostatitis, symptomatic prostatic hypertrophy, polycythemia, severe acne, breast cancer, prostate cancer, or hypopituitarism.
2. Currently being treated with testosterone.
3. Meets lifetime criteria for schizophrenia, schizoaffective disorder, any bipolar disorder (i.e., BP-I, BP-II, or BP NOS); or a major depressive episode in the preceding 5 years.
4. Current suicidal risk.
5. Current (past year) substance abuse or dependence.

Ages: 40 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Dates: Start 2004-09

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-d)
Clinical Global Impression- Change (CGI-C)
Profile of Mood States (POMS)
Beck Depression Inventory (BDI)
Sheehan Disability Scale
Self Anchoring Scale (SAS)
Affective Balance Scale (ABS)
International Index of Erectile Function (IIEF)
Aging Male Symptom rating (AMS)
Clinical Global Impression (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Orr, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Psychiatric out patient clinical unit, Tel Litwinsky, Israel